CLINICAL TRIAL: NCT03892941
Title: Electric Pace-pitched Hearing Achieves Natural Tonotopy
Acronym: ELEPHANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL64874.068.18
Record Dates: First submitted 2019-03-20; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaged based fitting (Experimental): Mapping of the electrical input of the cochlear implant will be based on an individualized natural frequency alignment as estimated with imaging methods.
  Interventions: Device: Imaged based fitting
- Clinical routine (No Intervention): Mapping of the electrical input of the cochlear implant will be based on a one-size-fits-all, as is part of clinical routine.

INTERVENTIONS:
Device: Imaged based fitting — Mapping of the electrical input of the cochlear implant will be based on an individualized natural frequency alignment as estimated with imaging methods.
  Arms: Imaged based fitting

SUMMARY:
In search of the best possible outcome for the severe hearing impaired who have regained the ability to hear by means of a cochlear implant (CI), electrical stimulation and the information it carries should match as closely as possible to what the human brain naturally has evolved to cope with and learned to process instead of relying on plasticity to adapt to an induced mismatch. At the moment, however, CI's are fitted with a 'one size fits all' principle. This is known to cause a mismatch between the frequencies presented by the CI electrode array and the frequencies represented at the corresponding natural acoustic location in an individual cochlea. In this study it is hypothesized that an individual imaged based fitting that pursues natural hearing alignment and is implemented from the start of the rehabilitation process, will improve the individual outcomes of electric hearing. The natural fitting strategy is thought to give rise to a steeper learning curve, result in a better performance in challenging listening situations, improve sound quality, complement better with residual acoustic hearing in the contralateral ear and win the preference of CI-recipients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18y or older) and meeting the conventional Dutch CI criteria;
* Proficient speaker of Dutch language;
* Post-lingual onset of profound deafness (> 4 years of age);
* Subject receives an Advanced Bionics implant with Midscala electrode and an Advanced Bionics sound processor;
* Prepared to use study specific hearing aid (Phonak) for the duration of the study;
* Rehabilitation at MUMC+ for the first year after surgery regarding CI as well as HA;
* Active participation in trial related procedures such as daily randomization and regular testing.

Exclusion Criteria:

* Physical or non-physical contraindications for MRI or CT imaging;
* Additional disabilities that may prevent active participation and testing as per protocol. If there are indications that the mental abilities to comply with the study procedures are insufficient, additional screening will be performed with the Mini-Mental State Examination. Patients will be excluded from the study when the resulting score is lower than 24;
* Cochlear or neural abnormalities that could affect outcome measures and/or compromise the placement of the electrode as assessed by the CI surgeon;
* Active participation in another prospective clinical trial;
* Pregnancy at time of imaging;
* Requirement for electric-acoustic activation prior to the first year follow-up;
* Having received a cochlear implant earlier (e.g. explantation or bilateral implantation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-03-18 (Estimated); Study Completion 2021-03-18 (Estimated)

PRIMARY OUTCOMES:
Speech understanding in quiet with cochlear implant | During the first 12 months of CI rehabilitation
  Speech understanding with CI in quiet measured with the Dutch Consonant Nucleus Consonant (CNC) test.
Speech understanding in quiet with cochlear implant | During the first 12 months of CI rehabilitation
  Speech understanding with CI in quiet will be measured with the Dutch Matrix sentence test.
Speech understanding in noise with cochlear implant | During the first 12 months of CI rehabilitation
  Speech understanding with CI in noise will be measured with the Dutch Matrix sentence test.
Patient preference | During the first 12 months of CI rehabilitation
  At every fitting session, patients will be asked to rate their satisfaction with either the control or experimental program on a 10-point Visual Analog Sscale (1 dissatisfied - 10 very satisfied).

SECONDARY OUTCOMES:
Speech understanding with hearing aid | During the first 12 months of CI rehabilitation
  Speech understanding with hearing aid will be measured with the Dutch Consonant Nucleus Consonant (CNC) test.
Speech understanding with hearing aid | During the first 12 months of CI rehabilitation
  Speech understanding with hearing aid will be measured with the Dutch Matrix sentence test.
Spatial masking | During the first 12 months of CI rehabilitation
  The Spatial Speech Perception In Noise (SSPIN) test will be used to determine the head shadow and squelch effect [74].
Listening effort | During the first 12 months of CI rehabilitation
  In a listening effort test subjects are asked to rate the effort it takes to listen to speech fragments in noise.The listening effort test is based on subjective ratings for the ease or difficulty involved in listening to speech in the presence of varying amounts of noise. Speech and noise are presented from the same loudspeaker in front of the subject. Three relevant signal-to noise ratios will be tested repeatedly (5 times) and the mean effort level will be calculated. Rating is performed using a vertical scale with 13 discrete points (seven named categories interspersed with an empty category) ranging from no effort (Score 0) to extreme effort (Score 12).
Spectral resolution (SMRT test) | During the first 12 months of CI rehabilitation
  The ability to spectrally resolve frequency information is known to be related to speech understanding performance (in noise). Frequency selectivity will be monitored to test the ability of the patient to filter out one stimulus from the others on the basis of frequency. This will be done with the Spectral-temporally Modulated Ripple Test (SMRT).
Loudness scaling (ACALOS test) | During the first 12 months of CI rehabilitation
  To estimate the course of loudness percept between minimal audible level and maximum comfortable level, a procedure is used that automatically adjusts the presentation levels to the subject's individual auditory dynamic range without employing any pre-measurement. The procedure uses repeated measurements and presents levels in randomized order. It has been named "ACALOS" (Adaptive Categorical LOudness Scaling). Results will provide information about the difference in loudness percept between CI and HA and will give input for optimizing the fitting of these hearing devices across the dynamic range.
Telemetric data | During the first 12 months of CI rehabilitation
  By measuring Evoked Compound Action Potential (ECAP), telemetric data on the function of the implant and the response of the auditory nerve will be collected.
Quality of life in relation to hearing ability. | During the first 12 months of CI rehabilitation
  Measured with the Speech-Spatial-Qualities (SSQ) questionnaire. A short form of the SSQ (SSQ-12) will be used. The SSQ is designed for use typically as a complement to behavioural or experimental measures of hearing ability and consists of questions on the following domains: speech hearing, spatial hearing, qualities of hearing, and listening effort. Participants will be asked to answer 12 questions on a 10-point Visual Analogue Scale with different units.
Overall wellbeing | During the first 12 months of CI rehabilitation
  Measured with the ICEpop CAPability measure for adults (ICECAP-A)
Overall Quality of life | During the first 12 months of CI rehabilitation
  Measured with the Health Utility Index Mark 3 (HUI-3)

CONTACTS AND LOCATIONS:
Overall Officials: Erwin George, Dr., Principal Investigator — Maastricht UMC
Locations (1):
- MUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lambriks LJG, van Hoof M, Debruyne JA, Janssen M, Chalupper J, van der Heijden KA, Hof JR, Hellingman CA, George ELJ, Devocht EMJ. Evaluating hearing performance with cochlear implants within the same patient using daily randomization and imaging-based fitting - The ELEPHANT study. Trials. 2020 Jun 23;21(1):564. doi: 10.1186/s13063-020-04469-x. PMID 32576247